CLINICAL TRIAL: NCT06981858
Title: A Single-Arm Exploratory Study of Enlansibumab Sequentially Combined With Concurrent Chemoradiotherapy for Locally Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZLS2025107-A
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: LOCALLY ADVANCED CERVICAL CANCERS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential Enlonstobart Injection with concurrent chemoradiotherapy (Experimental)
  Interventions: Drug: Enlonstobart Injection

INTERVENTIONS:
Drug: Enlonstobart Injection — Sequential Enlonstobart Injection with concurrent chemoradiotherapy

SUMMARY:
This is a prospective , single - arm clinical study , aiming to evaluate the efficacy and safety of Enlansibumab sequential concurrent chemoradiotherapy in locally advanced cervical cancer. Patients will first receive one cycle of Enlansibumab monotherapy (360 mg, 60 - min IV infusion on day 1, every 3 weeks). After one treatment cycle (3 weeks), they'll undergo imaging assessment. Then, they'll have Enlansibumab (360 mg, 60 - min IV infusion on day 1, every 3 weeks for two cycles) combined with concurrent chemoradiotherapy. Chemotherapy involves cisplatin (40 mg/m²) or carboplatin (AUC2) via IV infusion, weekly (±7 days), with five planned cycles. Investigators may add a sixth platinum - based chemotherapy cycle if needed. Radiotherapy comprises EBRT and BT and must be completed within eight weeks of treatment initiation. The total prescription dose of EBRT combined with BT should have an EQD2 of ≥8000 cGy, with adjustments based on tumor regression. After concurrent chemoradiotherapy, treatment ends. An imaging assessment occurs around seven days (±3 days) later. Then, the follow - up phase begins, including final, safety, and survival follow - ups, continuing until patients are lost to follow-up, the follow-up ends, or they die.

ELIGIBILITY:
Inclusion criteria:

1. Female, aged 18-70 years (including boundary values);
2. Diagnosed histologically as cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma; 3.2018 FIGO stage IIB-IVA; Assess lymph node involvement based on one of the following criteria:

   * Lymph node involvement confirmed by histology and biopsy;
   * MRI or CT shows one or more positive pelvic/abdominal aortic lymph nodes with a minimum diameter of ≥ 15mm;
   * PET/CT or PET/MR display one or more positive pelvic/abdominal aortic lymph nodes with SUVmax ≥ 2.5 and higher than the background value in surrounding normal tissues.

According to the evaluation criteria for solid tumor efficacy version 1.1 (RECIST v1.1), having at least one measurable lesion; 5.ECOG PS 0-1； 6. According to the researcher's judgment, those with an expected survival period of ≥ 3 months; 7. The subjects can provide tumor tissue sections to determine whether formalin fixed paraffin embedded tumor histopathological samples or fresh tumor histopathological samples can be used for PD-L1 expression and other immune indicators detection; 8. Have sufficient organ function and meet the following laboratory examination standards:

1. Blood routine (no blood transfusion within 14 days, no use of hematopoietic stimulating factors, and no use of other drugs to correct blood cell count): White blood cell count (WBC) ≥ 3000/mm3; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 90 × 109/L; hemoglobin (HGB) ≥ 9g/dL;
2. Blood biochemistry: creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN), if>1.5 × ULN, creatinine clearance rate must be ≥ 60mL/min, calculated using the Cockcroft Gault formula; Total bilirubin (TBIL) ≤ 1.5 × ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN;
3. Thyroid function: Thyroid stimulating hormone (TSH) ≤ ULN; If there are abnormalities, additional tests should be conducted on T3 and T4, and their levels should be normal; 9. Women of childbearing age who have a negative pregnancy test and are not breastfeeding, and have fertility, must receive effective medical contraception measures (from signing the informed consent form to within 6 months after the last study administration); 10. Participants must agree to collect blood samples, paraffin embedded (FFPE) tumor tissue specimens or sections, and fresh tumor tissue specimens for relevant research.

11. The subjects voluntarily participated in this study, had good compliance with the planned treatment and follow-up, understood the research process of this study, and voluntarily signed an informed consent form.

Exclusion criteria:

1. There are distant metastatic diseases present;
2. Have received any previous anti-tumor treatment, including but not limited to surgery (excluding biopsy), radiotherapy, or systemic therapy (chemotherapy, immunotherapy, targeted therapy);
3. Previous treatment with immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies;
4. Active malignant tumor within 3 years before the first administration, excluding cervical cancer studied in this trial and any locally curable tumor that has received radical treatment (such as excised basal cell or squamous cell skin cancer, superficial bladder cancer cancer or cured carcinoma in situ, such as breast carcinoma in situ);
5. Suffering from active autoimmune diseases, or having a history of autoimmune diseases within 2 years before enrollment, and still requiring systemic treatment. Autoimmune diseases include but are not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction, asthma requiring intervention with bronchodilators;
6. Suffering from primary immunodeficiency disease or having a medical history;
7. Individuals who have received immunosuppressive therapy (such as cyclosporine) or require systemic steroid therapy (such as>20 mg/day prednisone or equivalent) within the 14 days prior to enrollment, except for those who receive local corticosteroid therapy via nasal spray, inhalation, or other routes;
8. Individuals who are HIV Ab positive or have active syphilis infection; Hepatitis B virus surface antigen (HBsAg) is positive, and the detection value of hepatitis B virus is>500IU/ml or 2500 copies/mL; Hepatitis C antibody (HCV Ab) is positive, and the hepatitis C virus RNA quantification is greater than the upper limit of the normal value of the detection unit. (Note: For those with positive hepatitis B virus surface antigen (HBsAg), antiviral treatment is recommended before the first use of the study drug, and nucleoside analogs such as entecavir and tenofovir dipivoxil are recommended. )
9. Active bacterial, fungal, or viral infections (defined as requiring intravenous injection of antibacterial, antifungal, or antiviral drugs for treatment) within 14 days prior to enrollment. For individuals who have no clinical manifestations of active infection before the first medication and receive prophylactic treatment for infection, they may be considered for inclusion;
10. Active tuberculosis or medical history;
11. Have experienced severe cardiovascular disease within the 6 months prior to enrollment, including but not limited to: stable angina pectoris with functional classification of III-IV; Unstable angina or myocardial infarction; NYHA grade III-IV congestive heart failure; Severe arrhythmia requiring medication treatment (if ventricular rate can be controlled, asymptomatic atrial fibrillation subjects are allowed to be included); Serious arterial/venous thrombotic events (such as cerebral hemorrhage, cerebral infarction, deep vein thrombosis, and pulmonary embolism);
12. Suffering from uncontrollable hypertension;
13. Have previously suffered from interstitial lung disease or non infectious pneumonia requiring glucocorticoid treatment;
14. There is clinically significant hydronephrosis that cannot be relieved by nephrostomy or ureteral stent placement, as determined by researchers; Within 28 days prior to enrollment or planned to receive live or attenuated vaccine treatment during the study period;

16. Known recipients of organ transplantation or allogeneic hematopoietic stem cell transplantation; 17. Have a history of severe allergic reactions and uncontrolled allergic asthma to all components of monoclonal antibody preparations; 18. There are contraindications or severe allergic reactions to any component of cisplatin; 19. Individuals who have participated in other clinical trials and used the investigational drug within 28 days prior to enrollment; 20. Participants who may have poor compliance with the research procedures and requirements, as determined by the researchers, such as those with a clear history of neurological or psychiatric disorders (including epilepsy or dementia), current mental disorders, and substance abuse; 21. Individuals with a clear history of neurological or mental disorders or drug abuse who are unable to quit or have a history of drug use; 22. There are situations where other researchers have determined that it is not suitable to participate in this experiment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
1-year PFS rate | 1 year after treatment initiation

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol